CLINICAL TRIAL: NCT03218397
Title: Rapid Identification and Phenotypic Susceptibility Testing for Gram-Negative Bacteremia (RAPIDS-GN)
Brief Title: Rapid Identification and Phenotypic Susceptibility Testing for Gram-Negative Bacteremia
Acronym: RAPIDS-GN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00075768; 5UM1AI104681 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Gram-negative Bacteremia
Keywords: Gram-negative Bacteremia; ICU; Critically ill; Intensive Care Unit; Rapid identification; Rapid susceptibility; Accelerate PhenoTest™ BC Kit; Accelerate Pheno™ System (AXDX); Antimicrobial stewardship; Antimicrobial use
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Primary service/provider: The primary service, including the prescribing provider, will be unaware of group assignment at the time of randomization, so initial antibiotic choice will not be affected by group assignment. Once rapid results become available and/or AS interventions are made, treating providers may become aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard blood culture and AST (Active Comparator): Standard blood culture and antimicrobial susceptibility testing (AST), and antimicrobial stewardship.
  Interventions: Device: Standard Culture and AST
- Rapid organism identification and AST (Active Comparator): Rapid organism identification and AST using the Accelerate PhenoTest™ BC Kit, performed on the Accelerate Pheno™ System (AXDX), and antimicrobial stewardship. The blood sample will also undergo standard culture and AST in addition to the rapid testing.
  Interventions: Device: Accelerate PhenoTest™ BC Kit

INTERVENTIONS:
Device: Accelerate PhenoTest™ BC Kit — Rapid identification and AST using the Accelerate PhenoTest™ BC Kit, performed on the Accelerate Pheno™ System (AXDX)
  Arms: Rapid organism identification and AST
Device: Standard Culture and AST — Standard culture and antimicrobial susceptibility testing (AST)
  Arms: Standard blood culture and AST

SUMMARY:
RAPIDS-GN is a multi-center, prospective, randomized, controlled trial to evaluate the following strategies for patients with confirmed gram-negative bacillus bacteremia (GNB):

1. Standard culture and antimicrobial susceptibility testing (AST); or
2. Rapid identification and AST using the Accelerate PhenoTest™ BC Kit, performed on the Accelerate Pheno™ System (AXDX)

DETAILED DESCRIPTION:
RAPIDS-GN is a multi-center, prospective, randomized, controlled trial to evaluate the following strategies for patients with confirmed gram-negative bacillus bacteremia (GNB):

1. Standard culture and antimicrobial susceptibility testing (AST); or
2. Rapid identification and AST using the Accelerate PhenoTest™ BC Kit, performed on the Accelerate Pheno™ System (AXDX)

Patient specimens with positive blood culture with Gram stain showing GNB identified during local laboratory business hours will be enrolled by the Microbiology Laboratory Technologist if they do not meet any exclusion criteria. Subject specimens will be randomized 1:1 to standard culture and AST or Rapid identification and AST using the FDA approved Accelerate Pheno TM System. Both groups will receive standard antimicrobial stewardship (AS). The primary service, including the prescribing provider, will be unaware of group assignment at the time of randomization, so initial antibiotic choice will not be affected by group assignment. Once rapid results become available and/or AS interventions are made, treating providers may become aware of group assignment.

The goal of this study is to determine the impact of rapid bacterial identification and phenotypic antimicrobial susceptibility testing (AST) on antimicrobial usage and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Positive blood culture with Gram stain showing GNB identified during local laboratory business hours.

Exclusion Criteria:

* Identification of GNB outside of local laboratory business hours (e.g. whenever laboratories are staffed to perform both rapid testing and routine testing)
* Positive blood culture for GNB at the same institution within prior 7 days (if known at the time of randomization).
* Deceased at the time of randomization.
* GNB plus gram-positive organism, gram-negative cocci, and/or yeast detected on Gram stain
* Previous enrollment in this study
* No Minnesota research authorization (Rochester site only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Banerjee, MD, PhD, Study Chair — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee R, Komarow L, Virk A, Rajapakse N, Schuetz AN, Dylla B, Earley M, Lok J, Kohner P, Ihde S, Cole N, Hines L, Reed K, Garner OB, Chandrasekaran S, de St Maurice A, Kanatani M, Curello J, Arias R, Swearingen W, Doernberg SB, Patel R. Randomized Trial Evaluating Clinical Impact of RAPid IDentification and Susceptibility Testing for Gram-negative Bacteremia: RAPIDS-GN. Clin Infect Dis. 2021 Jul 1;73(1):e39-e46. doi: 10.1093/cid/ciaa528. PMID 32374822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Started | 249 | 251
Completed | 226 | 222
Not Completed | 23 | 29
Not completed — Prior positive blood culture | 8 | 13
Not completed — Comfort care | 8 | 5
Not completed — Comfort care and positive blood culture | 1 | 0
Not completed — Comfort care and mixed culture | 0 | 1
Not completed — Mixed culture | 2 | 2
Not completed — Inaccessible hospital records | 2 | 5
Not completed — No gram-negative bacilli (GNB) | 0 | 2
Not completed — Randomized during laboratory off hours | 2 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST | Total
Number analyzed (Participants) | 226 | 222 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (18.3) | 62.2 (20.3) | 64.0 (19.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 130 | 122 | 252
  Female | 95 | 100 | 195
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 29
  Not Hispanic or Latino | 202 | 191 | 393
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 9 | 8 | 17
  White | 183 | 176 | 359
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 21 | 26 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 226 | 222 | 448

OUTCOME MEASURES:

1. Primary Outcome: Hours to First Antibiotic Modification
Description: Mean hours until first modification of antibiotic therapy within 72 hours post randomization
Time Frame: 72 hours after randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 24.7 (24.6) | 19.0 (22.9)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.013, t-test, 2 sided — alpha = 0.05; Difference in means = 5.6, 95% CI 2-sided [1.2 to 10] — Difference in mean hours to first antibiotic modification (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

2. Secondary Outcome: Subjects Who Experienced Mortality Within 30 Days of Randomization
Description: Subjects who experienced mortality within 30 days of randomization
Time Frame: Within 30 days of randomization
Population: Subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
Participants
  Dead within 30 days | 18 | 25
  Not dead within 30 days | 206 | 197
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.265, Fisher Exact — alpha = 0.05

3. Secondary Outcome: Length of Stay in the Hospital
Description: Length of stay in the hospital after randomization, up to 30 days, for patients alive at 30 days. Length of stay will be date of discharge minus date of randomization.
Time Frame: Within 30 days of randomization
Population: Subjects who were alive at 30 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 208 | 197
days | 8.2 (8.7) | 9.8 (9.8)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.093, t-test, 2 sided — alpha = 0.05; T-test for the difference in mean length of stay (days) between treatment arms among subjects alive at 30 days

4. Secondary Outcome: ICU Status Through 72 Hours Post-randomization
Description: ICU status through 72 hours post-randomization
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
Participants
  In ICU < 72 hours after randomization | 33 | 55
  In ICU for >= 72 hours after randomization | 34 | 37
  Not in ICU | 159 | 130
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.014, Fisher Exact — alpha = 0.05

5. Secondary Outcome: Time to First Antibiotic Escalation
Description: Mean hours to first antibiotic escalation within 72 hours from randomization, where escalation is defined as changing to a broader spectrum antibiotic, addition of one or more antibiotics, or conversion of oral to intravenous route.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 52.7 (28.8) | 45.2 (31.4)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.009, t-test, 2 sided — alpha = 0.05; Difference in means = 7.5, 95% CI 2-sided [1.9 to 13.1] — Difference in mean hours to first antibiotic escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

6. Secondary Outcome: Time to First Gram-negative Antibiotic Escalation
Description: Mean hours to first gram-negative antibiotic escalation within 72 hours from randomization, where escalation is defined as changing to a broader spectrum antibiotic, addition of one or more antibiotics, or conversion of oral to intravenous route.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 53.9 (28.4) | 47.5 (31.2)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.022, t-test, 2 sided — alpha = 0.05; Difference in means = 6.5, 95% CI 2-sided [0.9 to 12.0] — Difference in mean hours to first gram-negative antibiotic escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

7. Secondary Outcome: Time to First Gram-positive Antibiotic Escalation
Description: Mean hours to first gram-positive antibiotic escalation within 72 hours from randomization, where escalation is defined as changing to a broader spectrum antibiotic, addition of one or more antibiotics, or conversion of oral to intravenous route.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 70.5 (9.5) | 69.7 (11.3)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.46, t-test, 2 sided — alpha = 0.05; Difference in means = 0.7, 95% CI 2-sided [-1.2 to 2.7] — Difference in mean hours to first gram-positive antibiotic escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

8. Secondary Outcome: Time to First Antibiotic De-escalation
Description: Mean hours to first antibiotic de-escalation within 72 hours from randomization, where de-escalation is defined as changing to a narrower spectrum antibiotic, cessation of one or more antibiotics, or changing from an intravenous to oral route of appropriate drug.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 44.2 (26.2) | 39.6 (28.0)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.074, t-test, 2 sided — alpha = 0.05; Difference in means = 4.6, 95% CI 2-sided [-0.4 to 9.6] — Difference in mean hours to first antibiotic de-escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

9. Secondary Outcome: Time to First Gram-negative Antibiotic De-escalation
Description: Mean hours to first gram-negative antibiotic de-escalation within 72 hours from randomization, where de-escalation is defined as changing to a narrower spectrum antibiotic, cessation of one or more antibiotics, or changing from an intravenous to oral route of appropriate drug.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 55.8 (23.5) | 49.3 (27.8)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.008, t-test, 2 sided — alpha = 0.05; Difference in means = 6.5, 95% CI 2-sided [1.7 to 11.2] — Difference in mean hours to first gram-negative antibiotic de-escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

10. Secondary Outcome: Time to First Gram-positive Antibiotic De-escalation
Description: Mean hours to first gram-positive antibiotic de-escalation within 72 hours from randomization, where de-escalation is defined as changing to a narrower spectrum antibiotic, cessation of one or more antibiotics, or changing from an intravenous to oral route of appropriate drug.
Time Frame: Within 72 hours of randomization
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
hours | 60.4 (22.6) | 62.2 (21.3)
Statistical Analysis 1: Comparison: Standard Blood Culture and AST vs Rapid Organism Identification and AST; Test type: Superiority; p = 0.37, t-test, 2 sided — alpha = 0.05; Difference in means = -1.9, 95% CI 2-sided [-5.9 to 2.2] — Difference in mean hours to first gram-positive antibiotic de-escalation (Standard Blood Culture and AST minus Rapid Organism Identification and AST)

11. Secondary Outcome: Number of Hospital-onset Clostridium Difficile Infections
Description: Acquisition of hospital-onset Clostridium difficile within 30 days, as defined by the National Healthcare Safety Network (NHSN), normalized to 10,000 patient-days.
Time Frame: Within 30 days of randomization
Population: Subjects who completed the study.
Measure: Number (95% Confidence Interval); unit: Infections per 10,000 patient-days
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
Infections per 10,000 patient-days | 26.8 [11.2 to 64.4] | 27.5 [12.4 to 61.3]

12. Secondary Outcome: Number of New Hospital-acquired Infections (HAIs) and/or Multidrug Resistant Organisms (MDROs), Normalized to 10,000 Patient-days.
Description: Acquisition of new hospital-acquired infections (HAIs) and/or multidrug resistant organisms (MDROs) within 30 days during index hospitalization identified on routine clinical or surveillance samples.
  Cultures that will be tracked include the following, from any specimen source, unless otherwise indicated:
  * Methicillin-resistant Staphylococcus aureus
  * Vancomycin-resistant Enterococcus
  * 3rd generation cephalosporin non-susceptible Enterobacteriaceae
  * Carbapenem-resistant Enterobacteriaceae, as defined by the Centers for Disease Control and Prevention (CDC): resistant to imipenem, meropenem, doripenem, or ertapenem OR documentation that the isolate possesses a carbapenemase
  * Multidrug-resistant Pseudomonas aeruginosa (resistant to aminoglycosides, cephalosporins, fluoroquinolones, and carbapenems)
  * Carbapenem-resistant Acinetobacter
  * Candida species (isolated from blood cultures only)
Time Frame: Within 30 days of randomization
Population: Subjects who completed the study.
Measure: Number (95% Confidence Interval); unit: Infections per 10,000 patient-days
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
Number analyzed (Participants) | 226 | 222
Infections per 10,000 patient-days | 123.3 [82.0 to 185.6] | 105.5 [70.1 to 158.8]

ADVERSE EVENTS:
Time Frame: 30 days from randomization
Description: With the exception of mortality, adverse events were not collected.
Arm/Group | Standard Blood Culture and AST | Rapid Organism Identification and AST
All-Cause Mortality (participants affected / at risk) | 18/226 | 25/222
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03218397/Prot_SAP_000.pdf